CLINICAL TRIAL: NCT06373822
Title: New Perspectives in Adenomyosis Pathogenesis With Epigenetic Analysis and miRNAs
Acronym: ADENO-MIRNA
Status: Recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/18JAN/028
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group (N=25): Female patients visiting the service de Gynécologie of the CUSL for the purpose of intervention in the context of a benign gynecological issue (myomectomy, endometrial resection etc).
  * Age ≥ 18 years
  * Pre-menopausal
  * Not HIV or Hepatitis-positive
  * Not having participated in another clinical study in the 12 months prior to recruitment
  * Not presenting symptoms of adenomyosis and/or endometriosis
  Interventions: Diagnostic Test: Circulating-mirna
- Adenomyosis group (N=25): Female patients visiting the service de Gynécologie of the CUSL for the purpose of surgical intervention in the context of uterine adenomyosis.
  * Age ≥ 18 years
  * Pre-menopausal
  * Not HIV or Hepatitis-positive
  * Not having participated in another clinical study in the 12 months prior to recruitment
  * Not presenting symptoms of endometriosis
  Interventions: Diagnostic Test: Circulating-mirna

INTERVENTIONS:
Diagnostic Test: Circulating-mirna — A single blood sample (1 tube of 10 ml) on the day of the patient's visit to the service de Gynécologie of the CUSL.

SUMMARY:
Objectives:

To identify differentially expressed miRNAs in the blood of adenomyosis patients in view to develop new diagnostic methods

Hypotheses Circulating miRNAs may be abnormally expressed in patients suffering from adenomyosis and could be used to diagnose the disease

Study Design Blood samples will be collected from healthy subjects and adenomyosis patients and miRNAs will be isolated and analyzed to detect potential differences.

DETAILED DESCRIPTION:
The present study is based on previous research pointing out that circulating miRNAs are abnormally expressed in several pathologies including endometriosis, and can be used as a handy diagnostic tool in the clinical setting. The investigators hypothesize that miRNAs are differentially expressed in adenomyosis as well and could serve as noninvasive biomarkers to diagnose the condition. To test this hypothesis, the investigators plan to conduct a pilot study on 50 patients (25 adenomyosis patients and 25 healthy subjects), in order to compare expression of different miRNAs between the groups and determine a suitable diagnostic panel. There is approximatively 25 women undergoing hysterectomy for adenomyosis over the course of a year at the CUSL. It is also a necessary population in order to obtain statistically analyzable datas. This panel may be tested in the future in a larger population for validation purposes.

Blood samples (10 ml) will be collected the day of the surgery by the anesthetist from female patients visiting the CUSL for the purpose of hysterectomy. Patients will be subdivided into two groups, namely the study group (n=25) including patients diagnosed with adenomyosis by MRI and/or ultrasonography prior surgery and the control group (n=25) consisting of patients with pathologies unrelated to the endometrium. After samples registration in CUSL biobank, they will be transferred to the research laboratory and serum will be collected immediately by centrifuging at 2500 rpm for 15 min at 4° C followed by storage at -80°C until further use. To isolate circulating miRNAs, a commercial kit (Qiagen miRNeasy serum/plasma kit) will be used and cDNA will be then synthesized using appropriate kit (Qiagen miScript II RT). Commercial miRNA arrays will be used to simultaneously quantify expression of around 1000 miRNAs and compare their expression profiles between adenomyosis patients and unaffected subjects. Individual RT-qPCR reactions will be then conducted to validate the results. Differentially expressed microRNAs in adenomyosis will be further analyzed to determine their target genes and subsequent affected biological functions, using appropriate databases (TargetScan and miRTarBase). This experimental approach will allow us to identify abnormally expressed miRNAs in adenomyosis compared to disease-free women. These can then be used as noninvasive biomarkers of the pathology and/or targeted for development of new therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Pre-menopausal

Exclusion Criteria:

* HIV or Hepatitis-positive
* having participated in another clinical study in the 12 months prior to recruitment
* presenting symptoms of endometriosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients visiting the service de Gynécologie of the CUSL for the purpose of surgical intervention in the context of uterine adenomyosis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2031-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Circulating-miRNA as diagnostic biomarkers | Throughout the entire study, aproximately during 6,5 years
  Sequencing miRNA

CONTACTS AND LOCATIONS:
Locations (1):
- CUSL, Brussels, Woluwe-Saint-Lambert, Belgium

IPD SHARING:
Plan to Share IPD: No